CLINICAL TRIAL: NCT05171270
Title: How Does PsAID Implementation Affect Treatment Intensification and Patient Satisfaction in PsA
Brief Title: AsseSSing Impact in pSoriatic Treatment
Acronym: ASSIST
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 287039
Record Dates: First submitted 2021-11-24; First posted 2021-12-28 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2023-12

CONDITIONS: Psoriatic Arthritis
Keywords: Treatment decisions; Impact of disease
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Psoriatic arthritis: Psoriatic arthritis Impact of Disease questionnaires (PsAID) used within routine clinic consultation.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — PsAID questionnaire

SUMMARY:
Psoriatic arthritis (PsA) is a form of inflammatory arthritis associated with the skin condition psoriasis. A variety of different treatments are used to try to control arthritis and skin psoriasis and management often involves trial and error to find the right medication for the right person. Very little is known about the decisions made to increase treatment in individual patients. Previous research in rheumatoid arthritis found that clinical measures of disease activity, patient reported outcomes and characteristics of the treating doctor all influenced the decision to change therapy in routine practice.

This investigators particularly want to establish whether routine use of the psoriatic arthritis impact of disease (PsAID-12) questionnaire in the clinic setting can enable a better understanding of the impact of PsA on each individual, improve physician-patient communication and lead to appropriate interventions. The PsAID-12 questionnaire is a relatively new European developed questionnaire measuring patient impact across 12 different domains in PsA.

This study will use routine implementation of the PsAID-12 questionnaire and see if this is related to treatment decisions and patient satisfaction. The investigators will also examine other factors that may influence treatment decisions including patient characteristics, physician characteristics, disease activity and quality of patient-physician interactions.

DETAILED DESCRIPTION:
This is an observational, cross-sectional study addressing the factors influencing treatment decisions in patients with PsA. Participants will be treated as usual in their routine clinical practice, but decisions on treatment will be recorded - whether treatment is escalated, unchanged or reduced, and why.

The study will be conducted in 25 rheumatology centres in Europe (UK, France, Germany, Spain and Italy) with five centres in each country. Each participant will only attend for one single study visit which is likely to last around 30 minutes in total. This will be alongside the participant's routine clinic visit. The PsAID-12 questionnaire will be implemented on a tablet computer but the remaining outcomes will be collected on paper CRFs and transferred to a database for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study and complete questionnaires in the local language.
* Aged 18 years or above.
* Diagnosed with PsA according to the ClASification of Psoriatic ARthritis (CASPAR) criteria and diagnosis confirmed by a rheumatologist (Taylor 2006).

Exclusion Criteria:

* Patients who don't speak or read the local language
* Patients who are not comfortable filling in an app-based questionnaire or paper CRF.
* Patients with a new diagnosis of PsA at the current clinic visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with a diagnosis of PsA
Sampling Method: Non-Probability Sample
Enrollment: 503 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-03-22 (Actual); Study Completion 2022-03-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- France (5):
  - CHU Gabriel-Montpied, Clermont-Ferrand
  - Centre Hospitalier Le Mans, Le Mans
  - Hopitaux Universitaires de Marseille, Marseille
  - GERPAL, Hopital de la Pitie, Paris
  - Centre Hospitalier Universitaire (CHU) de Toulouse, Toulouse
- Germany (5):
  - Klinikum Bamburg, Bamberg
  - Rheumatologische Schwerpunktpraxis, Berlin
  - Universitatsklinik Frankfurt, Frankfurt
  - Universitätsklinikum der Ruhr-Universität Bochum, Herne
  - MVZ für Rheumatologie Dr. Martin Welcker GmbH, Planegg
- Ospedale Regionale Cardarelli, Campobasso, Italy
- Spain (5):
  - Complejo Universitario de a Coruña, A Coruña
  - Hospital Clinic (Barcelona), Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario de Salamanca, Salamanca
- United Kingdom (5):
  - Manchester University NHS Foundation Trust, Manchester, Greater Manchester
  - Oxford University Hospital NHS Foundation Trust, Oxford, Oxfordshire
  - Midlands Partnership NHS Foundation Trust, Stafford, Staffordshire
  - Cardiff and Vale University LHB, Cardiff, Wales
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford, Yorkshire

IPD SHARING:
Plan to Share IPD: Undecided
Available on reasonable request

REFERENCES:
- [Derived] Watson L, Coyle C, Whately-Smith C, Brooke M, Kiltz U, Lubrano E, Queiro R, Trigos D, Brandt-Juergens J, Choy E, D'Angelo S, Delle Sedie A, Dernis E, Guis S, Helliwell P, Ho P, Hueber AJ, Joven B, Koehm M, Montilla C, Packham J, Pinto Tasende JA, Ramirez Garcia FJ, Ruyssen-Witrand A, Scrivo R, Twigg S, Soubrier M, Wirth T, Gossec L, Coates LC. An international multicentre analysis of current prescribing practices and shared decision-making in psoriatic arthritis. Rheumatology (Oxford). 2024 Dec 1;63(12):3449-3456. doi: 10.1093/rheumatology/kead621. PMID 38011669

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment in rheumatology outpatient clinics at sites between 12/07/2021 and 22/03/2022
Period: Overall Study
Arm/Group | Psoriatic Arthritis
Started | 503 (Over-recruitment due to errors at sites)
Completed (Over-recruitment due to errors at sites) | 503
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full population
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 503
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 247
  Male | 256
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 107
  Italy | 84
  France | 100
  Germany | 101
  Spain | 111

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Undergoing Treatment Escalation
Description: Treatment escalation definition includes increase in dose, frequency, change of route, new medication
Time Frame: During the consultation visit (around 30-60 mins)
Population: Full population
Measure: Count of Participants; unit: Participants
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 503
Participants | 160

2. Secondary Outcome: Number of Patients Undergoing Reduction of Therapy
Description: Treatment reduction definition includes decrease in dose, frequency, change in route, stopping medication
Time Frame: During the consultation visit (around 30-60 mins)
Population: Full population
Measure: Count of Participants; unit: Participants
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 503
Participants | 22

3. Secondary Outcome: Mean PsAID-12 Scores
Description: PsA impact of disease score (scale 0-10 where higher score is worse)
Time Frame: During the consultation visit (around 30-60 mins)
Population: Full population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 503
score on a scale | 3.6 (2.5)

4. Secondary Outcome: Median CollaboRATE Score
Description: Patient satisfaction with consultation (scale 0-9 where higher score is better)
Time Frame: During the consultation visit (around 30-60 mins)
Population: Full population
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 503
score on a scale | 9 [0 to 9]

5. Secondary Outcome: Median Perceived Efficacy on Patient-physician Interaction Score (PEPPI)
Description: A patient-reported questionnaire to assess their perceived efficacy in a healthcare consultation. This consists of 5 questions which the patient rates on a likert scale of 1 to 5. The score for each of the questions are summed together giving a score range of 5-25 where higher score is better)
Time Frame: During the consultation visit (around 30-60 mins)
Population: Full population
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 503
score on a scale | 23 [9 to 25]

6. Secondary Outcome: Median Score for Physicians Opinion of How PsAID 12 Influenced Treatment Decision
Description: Likert scale 1-5 where
  1. A lot more likely to decrease or not change therapy
  2. Somewhat more likely to decrease or not change therapy
  3. No impact on treatment decision
  4. Somewhat more likely to increase therapy
  5. A lot more likely to increase therapy A higher score means that the PsAID 12 was more likely to influence treatment decisions.
Time Frame: During the consultation visit (around 30-60 mins)
Population: Complete data
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Psoriatic Arthritis
Number analyzed (Participants) | 503
score on a scale | 3 [1 to 5]

ADVERSE EVENTS:
Time Frame: Single visit (1 hour)
Description: Standard definitions
Arm/Group | Psoriatic Arthritis
All-Cause Mortality (participants affected / at risk) | 0/503
Serious Adverse Events (participants affected / at risk) | 0/503
Other Adverse Events (participants affected / at risk) | 0/503

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT05171270/Prot_SAP_000.pdf